CLINICAL TRIAL: NCT07119905
Title: Association Between Matrix Metalloproteinase-9 Gene Polymorphism and Susceptibility to Primary Open Angle Glaucoma Patients in Sohag University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Thomas Talaat Nageh, Demonstrator, Sohag University
Other Study IDs: Soh-Med--25-7-16MS
Record Dates: First submitted 2025-08-02; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: Primary Open Angle Glaucoma; POAG; Gene Polymorphism; MMP-9; Matrix Metalloproteinase-9 Gene Polymorphism
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Normal healthy volunteers aged > 30 years
  Interventions: Genetic: genotyping assay by polymerase chain reaction
- Experimental Group: Patients aged >30 years and diagnosed with Primary Open Angle Glaucoma
  Interventions: Genetic: genotyping assay by polymerase chain reaction

INTERVENTIONS:
Genetic: genotyping assay by polymerase chain reaction — Blood sample will be obtained from all participants by withdrawing 3 mL of blood via venipuncture in ethylenediaminetetraacetic acid tube.
  Thereafter, DNA extraction will be obtained after centrifugation to be used for genotyping assay of MMP-9 gene with polymerase chain reaction

SUMMARY:
The goal of this observational study is to investigate the potential association between MMP-9 gene polymorphism and susceptibility to Primary Open Angle Glaucoma development in Egyptian patients The main question it aims to

DETAILED DESCRIPTION:
Glaucoma is the second most common cause of blindness worldwide. Glaucoma is a progressive optic neuropathy, characterized by a specific loss of retinal nerve fibres and ganglion cells, gradual decrease of the visual ﬁeld, and vertical elongation of optic disc cupping. Glaucoma causes a slow loss of vision in the centre of the field of view as well as in the periphery. This results in delays in the diagnosis and treatment, and it is likely that the glaucoma may not be diagnosed until the disease has progressed to a moderate or severe level, at which point significant vision loss will have already taken place

POAG is the most common type of glaucoma that is characterized by speciﬁc glaucomatous retinal, optic nerve, and clinical ﬁndings without a clear secondary cause.

POAG is a progressive optic neuropathy characterized by loss of ganglion cells and deterioration of the visual ﬁeld in eyes with gonioscopically open angles, either with or without increased intraocular pressure (IOP).

Matrix Metalloproteinase-9 gene Matrix metalloproteinases (MMPs) are a kind of calcium-zinc ion-dependent proteolytic enzyme involved in a variety of cellular processes. MMPs are well known for their ability to degrade the extracellular matrix (ECM) and are involved in several intracellular mechanisms from cell differentiation, proliferation, and angiogenesis to apoptosis.

The MMP genes were suggested to play an important role in the development of various glaucoma types, MMPs are important regulators of the aqueous humor outﬂow from the eye anterior chamber and therefore significantly affect intraocular pressure. Patients with diagnosed POAG have an altered MMPs level in the aqueous humor.

Several studies have been conducted to analyze polymorphic variants of the MMP for their possible contribution to POAG, Several loci of the MMP genes (rs3918242, rs3918249, rs17576 matrix metalloproteinase-9 were associated with POAG.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 30 years
* Primary open angle glaucoma as evidenced from characteristic visual field loss and optic disc cupping (POAG group)
* Healthy subjects matched by age, sex and ethnicity to the POAG patients group (control group)

Exclusion Criteria:

* Exfoliation glaucoma, pigmentary glaucoma
* History of acute angle closure

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Primary Open Angle Glaucoma in Department of ophthalmology in Sohag University Hospitals and healthy controls of matched age and sex
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Matrix metalloproteinase-9 gene polymorphism | 14 months
  Matrix metalloproteinase-9 gene polymorphism by polymerase chain reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hosipital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grzybowski A, Och M, Kanclerz P, Leffler C, Moraes CG. Primary Open Angle Glaucoma and Vascular Risk Factors: A Review of Population Based Studies from 1990 to 2019. J Clin Med. 2020 Mar 11;9(3):761. doi: 10.3390/jcm9030761. PMID 32168880
- [Background] Liu Y, Allingham RR. Major review: Molecular genetics of primary open-angle glaucoma. Exp Eye Res. 2017 Jul;160:62-84. doi: 10.1016/j.exer.2017.05.002. Epub 2017 May 10. PMID 28499933
- [Background] Zhao F, Fan Z, Huang X. Role of matrix metalloproteinase-9 gene polymorphisms in glaucoma: A hospital-based study in Chinese patients. J Clin Lab Anal. 2020 Mar;34(3):e23105. doi: 10.1002/jcla.23105. Epub 2019 Nov 12. PMID 31713905